CLINICAL TRIAL: NCT07099911
Title: Novel Use of Neuromuscular Electrical Stimulation to Improve Glucose Control in Individuals With Spinal Cord Injury
Brief Title: Neuromuscular Electrical Stimulation and Glucose Control in Spinal Cord Injury
Acronym: NMES-SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Collaborators: University of Birmingham (Other)
Responsible Party: Principal Investigator, Jennifer Maher, PhD Programme for Health, University of Bath
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 346844; SBF009\1017 (Other Grant/Funding Number: Academy of Medical Sciences)
Record Dates: First submitted 2025-07-15; First posted 2025-08-01 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Spinal Cord Injury
Keywords: Neuromuscular electrical stimulation; Spinal cord injury; Glucose control; Metabolism
MeSH Terms: conditions — Spinal Cord Injuries | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal Cord Injury (Experimental): Participants will undergo two 3-hour oral glucose tolerance tests (OGTTs) with dual stable isotope tracers in a randomized crossover design. One OGTT will be paired with an acute bout of neuromuscular electrical stimulation (NMES), and the other with a sham condition (SHAM). After the OGTT sessions, participants will complete a 2-week period of at-home NMES use to assess real-world feasibility and acceptability through interviews.
  Interventions: Behavioral: NMES; Behavioral: Sham (No Treatment)
- Non-injured Control (CON) (Active Comparator): Age- and sex-matched individuals without SCI. Participants will undergo two 3-hour oral glucose tolerance tests (OGTTs) with dual stable isotope tracers in a randomized crossover design. One OGTT will be paired with an acute bout of NMES, and the other with a sham condition (SHAM). CON will not participate in the at-home NMES phase.
  Interventions: Behavioral: NMES; Behavioral: Sham (No Treatment)

INTERVENTIONS:
Behavioral: NMES — Acute bout of neuromuscular electrical stimulation during a 3-h OGTT.
Behavioral: Sham (No Treatment) — Sham stimulation during a 3-h OGTT.

SUMMARY:
Overall aim: To identify the impact and acceptability of a novel method of neuromuscular electrical stimulation (NMES) for improving glucose control using a dual stable isotope tracer OGTT in individuals with spinal cord injury (SCI).

Objective 1:

1. To establish the extent to which an acute bout of NMES improves health-related measures of glucose control, compared to a SHAM control trial.
2. To identify the relative magnitude of effect, compared to non-injured control participants (CON).

Hypotheses:

1. NMES will be more effective at improving glucose control by increasing peripheral glucose uptake, relative to SHAM condition.
2. The effect will be greater in individuals with SCI compared to non-injured control participants.

Objective 2:

To investigate the real-world feasibility of NMES as a therapeutic intervention, participants with SCI will be given instructions for 2-weeks of at-home use. In-depth interviews will be conducted to evaluate acceptability and identify areas that could be adapted to effectively implement NMES in a future trial.

Participants will complete two experimental trials in a randomised crossover fashion separated by 7 days which will consist of either a sham control (SHAM) or an acute bout of NMES during a 3-h oral glucose tolerance test (OGTT). Following the experimental trial days, participants with SCI will take home a NMES device and will be given instructions for 2-weeks of at-home NMES use (Figure 1) to assess acceptability and feasibility.

ELIGIBILITY:
Inclusion Criteria:

We are asking all individuals who meet our study criteria if they would like to take part. We are looking for both males and females who meet all the criteria on this list for either SCI or non-injured individuals:

Individuals with SCI:

* >1-year postinjury.
* 18 years of age or above
* American Spinal Cord Injury Impairment Scale A-C.
* Level of Injury, Cervical 5-Lumbar 2.
* Have capacity to provide informed consent.

Non-injured individuals:

• 18 years of age or above

Exclusion Criteria:

* Has been diagnosed with type 2 diabetes, or actively taking a pharmaceutical to address elevated blood glucose.
* Unable to understand explanations and/or provide informed consent.
* If you cannot tolerate the NMES intervention
* Is pregnant or planning to become pregnant during the study duration

SCI only:

* Recently trained with electrical stimulation (< 6 months)
* Recent history of lower limb fractures
* Peripheral nerve injury to lower extremities
* Unresolved pressure ulcers
* Known lower motor neuron injury.
* If the research team cannot induce visible or palpable contractions of the quadricep muscle with NMES
* If they cannot tolerate the NMES intervention
* Has previously experienced uncontrolled autonomic dysreflexia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-08 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Glucose incremental area under the curve (iAUC). | 180 minutes
  Glucose incremental area under the curve (iAUC) during oral glucose tolerance test (OGTT)
Glucose Kinetics | 0, 180 minutes post ingestion
  Glucose kinetics calculated from plasma deuterated glucose enrichment, including rate of appearance of endogenous glucose, rate of disappearance of glucose, and rate of appearance of exogenous glucose.

SECONDARY OUTCOMES:
Whole-body carbohydrate oxidation | 0,60,120,180 minutes post-ingestion
  Assessed via indirect calorimetry during 180-min OGTT (60-min intervals)
Whole body fat oxidation | 0, 60, 120, 180 minutes post-ingestion
  Assessed via indirect calorimetry during 180-min OGTT (60-min intervals)
Non-oxidative glucose disposal | 180 minutes
  Non-oxidative glucose disposal
Fasting plasma glucose concentration | Baseline
  Fasting plasma glucose concentration (mmol/L)
Fasting plasma non-esterified fatty acid concentrations | Baseline
  Fasting plasma non-esterified fatty acid concentrations (mmol/L)
Fasting plasma lactate concentrations | Baseline
  Fasting plasma lactate concentrations (mmol/L)
Postprandial non-esterified fatty acid concentrations | 15, 30, 45, 60, 90, 120, 150, 180 minutes post-ingestion
  Postprandial non-esterified fatty acid concentrations (mmol/L) in response to oral glucose tolerance test
Postprandial lactate concentrations | 15, 30, 45, 60, 90, 120, 150, 180 minutes post-ingestion
  Postprandial lactate concentrations (mmol/L) in response to OGTT
Total daily energy expenditure | 5 days
  Derived from indirect calorimetry and acccelerometry/heart rate monitoring.
Acceptability of at-home NMES | 2-weeks
  Acceptability of at-home NMES obtained via a survey and semi-structured interview.
Circulating endothelial cells | 0, 60, 120, 180 minutes post-ingestion of OGTT
  Circulating endothelial cells count/ml blood
Circulating endothelial progenitor cells | 0, 60, 120, 180 minutes post-ingestion of OGTT
  Circulating endothelial progenitor cell count/100 leukocytes
Tumor Necrosis Factor alpha (TNF-α) | 0, 60, 120, 180 minutes post-ingestion of OGTT
  Tumor Necrosis Factor alpha (TNF-α) (pg/mL)
Interleukin-6 (IL-6) | 0, 60, 120, 180 minutes post-ingestion of OGTT
  Interleukin-6 (IL-6) (pg/mL)
Interferon gamma (IFN-γ) | 0,60,120,180 minutes post-ingestion of OGTT
  Interferon gamma (IFN-γ) (pg/mL)

CONTACTS AND LOCATIONS:
Locations (1):
- Department for Health, University of Bath, Bath, United Kingdom, United Kingdom

IPD SHARING:
Plan to Share IPD: No